CLINICAL TRIAL: NCT00252746
Title: A Randomised, Double-blind, Parallel-group, Dose Finding Study to Assess the Efficacy and Safety of ZD6474 in Patients With Advanced, Metastatic, or Recurrent NSCLC Who Have Failed Previous Chemotherapy Regimens, at Least One of Which Contained Platinum [Title Abbreviated]
Brief Title: ZD6474 Phase IIa Dose Finding Multicentre Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4200C00039
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vandetanib

ARMS (3):
- ZD6474 100mg (Experimental): Daily dose
  Interventions: Drug: ZD6474 (vandetanib) 100mg
- ZD6474 200mg (Experimental): daily dose
  Interventions: Drug: ZD6474 (vandetanib) 200mg
- ZD6474 300mg (Experimental): daily dose
  Interventions: Drug: ZD6474 (vandetanib) 300mg

INTERVENTIONS:
Drug: ZD6474 (vandetanib) 100mg — once daily oral dose
  Other Names: ZACTIMA™
  Arms: ZD6474 100mg
Drug: ZD6474 (vandetanib) 200mg — once daily oral dose
  Other Names: ZACTIMA
  Arms: ZD6474 200mg
Drug: ZD6474 (vandetanib) 300mg — once daily oral dose
  Other Names: ZACTIMA
  Arms: ZD6474 300mg

SUMMARY:
To assess the objective response rates (by RECIST) to ZD6474 100, 200 and 300 mg/day respectively

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Life expectancy of 12 weeks or longer.

Exclusion Criteria:

* Pregnancy, breast feeding or female patients wishing to become pregnant.
* Treatment with a non-approved or investigational drug within 30 days before enrolment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To assess the objective response rates (by RECIST) to ZD6474 100, 200 and 300 mg/day respectively | Every 4 weeks for the first 24 weeks of treatment and then every 8 weeks until PD is determined or withdrawal due to any reasons other than PD. If PR or CR is observed, tumour assessment will be repeated 4 weeks after for confirmation of the response

SECONDARY OUTCOMES:
To assess the tolerability, safety, disease control rate, duration of response, time to progression, changes in quality of life and tumour-related and overall symptom improvements, and to characterise the PK and PK-PD relationship | Every 4 weeks till meeting discontinuation criteria
  Tumour assessments to evaluate disease control rate, duration of response, time to progression will be performed every 4 weeks for the first 24 weeks of treatment, then every 8 weeks until PD is determined or withdrawal due to any reasons other than PD. If PR or CR is observed, tumour assessment will be repeated 4 weeks after for confirmation of the response. Quality of life questionnaire - FACT-L will be given to subjects at baseline and at 4-week intervals during the study treatment (up to Week 12). Lung cancer subscale (LCS) for disease-related symptoms collection will be completed weekly (up to Week 12). Safety and tolerability will be assessed on the ongoing basis by AZ collection, and at the site visits by vital sign, ECG and lab assessments. Blood sampling for pharmacokinetics will be performed on day 8, 15, 22, 29, 57 and 85. In the event of QTc prolongation, PK sampling will continue with the additional ECG monitoring performed until the QTc has fallen below 460 msec.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Japan (7):
  - Research Site, Matsuyama, Ehime
  - Research Site, Isehara, Kanagawa
  - Research Site, Okayama, Okayama-ken
  - Research Site, Sayama, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Tokyo

REFERENCES:
- [Background] Kiura K, Nakagawa K, Shinkai T, Eguchi K, Ohe Y, Yamamoto N, Tsuboi M, Yokota S, Seto T, Jiang H, Nishio K, Saijo N, Fukuoka M. A randomized, double-blind, phase IIa dose-finding study of Vandetanib (ZD6474) in Japanese patients with non-small cell lung cancer. J Thorac Oncol. 2008 Apr;3(4):386-93. doi: 10.1097/JTO.0b013e318168d228. PMID 18379357